CLINICAL TRIAL: NCT01785121
Title: Increasing Exercise Capacity of Patients With Heart Failure by Wii Gaming (HF-Wii) A Randomized Controlled Trial
Brief Title: Increasing Exercise Capacity of Patients With Heart Failure by Wii Gaming
Acronym: HF-Wii
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: The Swedish Research Council (Other Government); The Swedish Heart and Lung Association (Other); Swedish Heart Lung Foundation (Other); Vardalinstitutet The Swedish Institute for Health Sciences (Other); Medical Research Council of Southeast Sweden (Other Government); Swedish Council for Working Life and Social Research (Other)
Responsible Party: Principal Investigator, Tiny Jaarsma, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HF-Wii
Record Dates: First submitted 2013-02-01; First posted 2013-02-07 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator): Patients who are randomized to the MSO group will get a protocoled exercise advice from a member of the HF team (nurse, cardiologist or physiotherapist). During the first three months after inclusion, patients will be phoned after 2, 4, 8, 12 weeks to discuss their current activity.
  Interventions: Behavioral: Motivational support only
- Wii Group (Experimental): Patients who are randomized to the Wii group will be introduced to the Nintendo Wii game computer in an introduction lesson of approximately two hours and the Wii will be installed at home. During the first three months after inclusion, patients will be phoned after 2, 4, 8, 12 weeks to discuss their experiences with the Wii or to solve possible problems
  Interventions: Behavioral: Structured access to a Wii game computer (Wii)

INTERVENTIONS:
Behavioral: Structured access to a Wii game computer (Wii) — Patients who are randomized to the Wii group will be introduced to the Nintendo Wii game computer in an introduction lesson of approximately two hours and the Wii will be installed at home. During the first three months after inclusion, patients will be phoned after 2, 4, 8, 12 weeks to discuss their experiences with the Wii or to solve possible problems
  Other Names: Wii group
  Arms: Wii Group
Behavioral: Motivational support only — The control group receives an protocolized exercise advice and telephone follow-up at 2, 4, 8 and 12 weeks
  Other Names: MOS
  Arms: Control Group

SUMMARY:
The study objectives are to determine the effectiveness of structured access to a Wii game computer compared to motivational support only in heart failure patients on exercise capacity and daily activity. Secondly, to determine the effectiveness of structured access to a Wii game computer compared to motivational support only in heart failure patients on the combined endpoint of death, readmission and quality of life.

The following research questions will be addressed:

* What is the effectiveness of structured introduction and access to a Wii game computer in patients with heart failure to improve their exercise capacity compared to patients with heart failure in a control group who only receive motivational support?
* What is the effectiveness of structured introduction and access to a Wii game computer in patients with heart failure compared to patients with heart failure in a control group who only receive motivational support to increase their daily physical activity, decrease health care use and improve quality of life?
* What are experiences of heart failure patients and how is their exercise motivation when they are introduced and instructed to play with a Wii game computer?

DETAILED DESCRIPTION:
Substudy

HF-WII PLUS MEDIYOGA

In this substudy Medical Yoga will be tested in a randomized group next to the Wii and the control group in the HF-Wii study and therefore the substudy will be called HF-Wii plus MediYoga.

In addition to the usual treatment and information about rehabilitation and daily activities for heart failure patients, this group will train a 60-minute yoga class twice a week. Patients will sit on chairs or yoga mats to perform yoga. Each patient will perform a total of 20-24 sessions over a 12-weeks period. A session will include 10 min warm-up and breathing exercises, 40 minutes of yoga postures and finally 10 min relaxation and meditation. At the end of each session, participants have the opportunity to discuss their experiences or questions. At the first visit, participants will receive a CD and a booklet with yoga postures and instructions. Patients are encouraged to train Medi Yoga at home with a target of one session a day. All yoga sessions will be conducted by a certified Medicare Yoga instructor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HF (NYHA I-IV) (independent of Ejection Fraction: both patients with a preserved ejection fraction (HFPEF) or reduced ejection fraction (HFREF) can be included)
* Older than 18 years, there is no upper age limit
* Speak/understand the language of the country where the intervention is taken place

Exclusion Criteria:

* The patient is expected to be unable to use the Nintendo Wii due to visual (see a TV screen at a distance of 3 m) cognitive (assessed by the HF nurse or cardiologist) or motor impairment (the patient should be able to swing his arm at least 10 times in a row)
* The patient has restrictions that would them unable patients to fill in data collection material
* The patient has a life expectancy shorter than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
change in 6 minute walk test | 3 months
  The 6 minute walk test measures the amount of meters covered by a patients in 6 minutes using a protocolled assessment

SECONDARY OUTCOMES:
Muscle function | Baseline, 3, 6, 12 months
  assessed with bilateral isometric shoulder abduction and unilateral isotonic shoulder flexion using predefined protocols
Exercise Motivation | Baseline, 3, 6, 12 months
  assessed by the Exercise motivation Index (EMI)
Daily Physical Activity | monitored every day during 6 months
  measured by an activity monitor
Exercise Self-Efficacy | Baseline, 3, 6, 12 months
  assessed by the exercise self-efficacy questionnaire (SEE)
Perceived Physical Effort | Daily for the first 3 months
  assessed with the Borg's scale of perceived exertion
Heart Failure Symptoms | Daily for the first 3 months
  assessed using a 10 point VAS scale
Health Related Quality of Life | Baseline, 3, 6, 12 months
  assessed with Minnesota Living with Heart Failure Questionnaire(MLWHFQ)
Global Well-Being | Daily for the first 3 months
  assessed with Cantril's ladder of life
Readmission | 12 months
  assessed from the medical record
Costs | 12 months
  cost of readmission, bed days occupancy (all cause) in medical/surgical beds, home care, contacts with and interventions of primary care, cost of the intervention (Wii game computer, instruction session etc.) and developing the intervention, materials and laboratory tests used
Experiences of patients | 12 months
  An open ended survey will be used to collect data on patient's experiences and challenges
change in 6 minute walk | 6 and 12 monhts

CONTACTS AND LOCATIONS:
Locations (10):
- University of California, Irvine, California, United States
- Center of Internal Medicine Elsterwerda, Elsterwerda, Germany
- Rabin Medical Center, Petah Tikva, Israel
- Villa delle Querce hospital, Nemi, Italy
- Maastricht University Medical Center, Maastricht, Netherlands
- Sweden (5):
  - Länssjukhuset Ryhov hospital, Jönköping
  - University hospital Linköping, Linköping
  - Vrinnevi Hospital, Norrköping
  - Nyköpings lasarett hospital, Nyköping
  - Karolinska University Hospital Huddinge, Stockholm

REFERENCES:
- [Derived] Klompstra L, Hagglund E, Jaarsma T, Kato NP, Stromberg A. Effects of exergaming and yoga on exercise capacity and physical and mental health in heart failure patients: a randomized sub-study. Eur J Cardiovasc Nurs. 2025 Apr 11;24(3):389-398. doi: 10.1093/eurjcn/zvae155. PMID 39743240
- [Derived] Klompstra L, Mourad G, Jaarsma T, Stromberg A, Alwin J. Costs of an Off-the-Shelf Exergame Intervention in Patients with Heart Failure. Games Health J. 2023 Jun;12(3):242-248. doi: 10.1089/g4h.2022.0013. Epub 2022 Dec 5. PMID 36473172
- [Derived] Poli A, Kelfve S, Klompstra L, Stromberg A, Jaarsma T, Motel-Klingebiel A. Prediction of (Non)Participation of Older People in Digital Health Research: Exergame Intervention Study. J Med Internet Res. 2020 Jun 5;22(6):e17884. doi: 10.2196/17884. PMID 32501275
- [Derived] Jaarsma T, Klompstra L, Ben Gal T, Ben Avraham B, Boyne J, Back M, Chiala O, Dickstein K, Evangelista L, Hagenow A, Hoes AW, Hagglund E, Piepoli MF, Vellone E, Zuithoff NPA, Martensson J, Stromberg A. Effects of exergaming on exercise capacity in patients with heart failure: results of an international multicentre randomized controlled trial. Eur J Heart Fail. 2021 Jan;23(1):114-124. doi: 10.1002/ejhf.1754. Epub 2020 Mar 13. PMID 32167657
- [Derived] Jaarsma T, Klompstra L, Ben Gal T, Boyne J, Vellone E, Back M, Dickstein K, Fridlund B, Hoes A, Piepoli MF, Chiala O, Martensson J, Stromberg A. Increasing exercise capacity and quality of life of patients with heart failure through Wii gaming: the rationale, design and methodology of the HF-Wii study; a multicentre randomized controlled trial. Eur J Heart Fail. 2015 Jul;17(7):743-8. doi: 10.1002/ejhf.305. PMID 26139585